CLINICAL TRIAL: NCT06274190
Title: Towards Personalized Care Pathways for Bowel Symptoms in Rectal Cancer Patients Through Precision Medicine
Brief Title: Personalized Care Pathways for Bowel Symptoms in Rectal Cancer patients_development of E-diary
Acronym: Treatable
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Inge Geraerts, Professor Dr., KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S68746
Record Dates: First submitted 2024-01-31; First posted 2024-02-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer; LARS - Low Anterior Resection Syndrome
Keywords: Bowel diary; Quality of Life (QoL); Care pathway
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Pre-Delphi patient focus group (No Intervention): During this focus group, we aim to achieve various goals:
  * To gain insight into the bowel symptoms and the consequences patients experienced after treating rectal cancer
  * To understand the expectations of the patients regarding an electronic bowel diary
  * To determine whether the questions/items derived from the literature study for the bowel diary are clear and understandable for the patients
  * To explore other relevant questions/items that should be added to the bowel diary
  We will include 8-12 patients in this focus group.
- Delphi survey (No Intervention): In this Delphi survey, a multidisciplinary group of experts and patients will score each item of the long list on a 1-9-point Likert scale from 'Not relevant' (1) to 'Essential' (9) for inclusion in the bowel diary. Finally, a patient consultation meeting and a consensus meeting will be held for the participants who completed the Delphi survey.
  We will recruit 10-18 Delphi panelists per area of expertise. These panelists are experts with international expert recognition in treating bowel symptoms in the following health care categories (abdominal surgeons, digestive/radiation oncologists, specialized pelvic floor muscle physiotherapists, nursing specialists). In addition, we will include one group comprising 10-18 patients in the Delphi survey, ensuring a comprehensive and holistic perspective on treating bowel symptoms across various healthcare categories.
- Post-Delphi patient focus group (No Intervention): During this focus group, our objective is to ensure that both the questions and answers are meaningful.
  We will include 8-12 patients in this focus group.
- Usability of e-diary (Experimental): The participants will be asked to use the newly developed electronic bowel diary for 7 consecutive days.
  To evaluate the usability of the e-diary, a group of 10 patients will participate in the assessment using the System Usability Scale (SUS).
  Furthermore we will have conversations with these patients regarding the use of the application: complexity, need for additional support, coherence of the application, user-friendliness, and the need for prior knowledge.
  Interventions: Diagnostic Test: bowel e-diary
- Psychometric properties of e-diary (Experimental): To evaluate the validity of the e-diary, encompassing test-retest reliability, construct validity and responsiveness, participants will be instructed to use the e-diary for two separate 7-day periods.
  Interventions: Diagnostic Test: bowel e-diary

INTERVENTIONS:
Diagnostic Test: bowel e-diary — This bowel diary will be available on the smartphone in the form of an application.
  Arms: Psychometric properties of e-diary; Usability of e-diary

SUMMARY:
Colorectal cancer is the 2nd and 3rd most common cancer in respectively women and men, of which about 40% is located in the rectum. The gold standard treatment for rectal cancer (RC) is a low anterior resection, combined with chemoradiotherapy. However, this treatment will negatively impact different aspects of bowel function and the patients' quality of life. These bowel symptoms often remain prevalent, even at 12 months after RC treatment. Most assessment tools are however not capable of capturing the full range or therapeutic-related evolution of these bowel symptoms. Consequently, the aim is to develop a validated bowel diary for diagnosing and evaluation of all bowel symptoms.

DETAILED DESCRIPTION:
Colorectal cancer is the 2nd and 3rd most common cancer in women and men, respectively and represents approximately 13% of all new cancer diagnoses, with 40% of cases specifically situated in the rectum. The gold standard treatment for rectal cancer (RC) is a low anterior resection, combined with chemoradiotherapy. However, given the improved oncological results, functional outcomes, such as bowel symptoms, become more and more important. Approximately 60-90% of RC patients are affected with a wide range of new onset bowel symptoms (incontinence for flatus or feces (solid, liquid), frequent bowel movements, urgency, clustering of defecation and evacuation problems) immediately after rectal treatment. The combination of these specific bowel symptoms and their impact on quality of life (QoL) has been summarized in an international consensus definition and is referred to as the Low Anterior Resection Syndrome (LARS).

Major LARS has an important impact on QoL and has major health economic consequences. This is attributable to its high prevalence after RC treatment, the chronic nature of symptoms and the limited evidence of available therapeutic options. This context leads to repetitive medical consultations, additional technical examinations which are often not very useful and need for prolonged medical treatment (multiple drug regimens), with often limited therapeutic gain. Furthermore, there is a lack of a comprehensive scoring system to identify the different aspects of LARS, leading to inadequate diagnostics and follow-up of symptoms. Based on these considerations, there is a clear need for a comprehensive scoring system for identification of the different aspects of LARS and monitoring of therapeutic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
* At least 18 years of age at the time of signing the Informed Consent Form (ICF).
* Proficient in reading, comprehending, and conversing in Dutch .
* Patients diagnosed with a rectal tumour based on a pathology report.

Exclusion Criteria:

* The participant has undergone a different type of surgery, including a Hartmann procedure, abdominoperineal excision, transanal endoscopic microsurgery, or sigmoid resection.
* Experienced fecal incontinence prior to undergoing surgery.
* Are affected by neurological disorders affecting bowel function.
* Already underwent previous pelvic surgery, previous pelvic radiation or rectal surgery for non-cancer reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2025-08-17 (Actual)

PRIMARY OUTCOMES:
Selection of items for the newly developed bowel diary | 12 months
  The selection of items for a comprehensive bowel diary in patients with rectal cancer is based on a literature review, a patient focus group and an international Delphi survey. The patient focus group is recorded using an audio and video recording. This recording is transcribed verbatim by the researcher into a Word document. The transcription will be analyzed using NVIVO 9 software. In this Delphi survey, a multidisciplinary group of experts will score each item of the long list on a 1-9-point Likert scale from 'Not relevant' (1) to 'Essential' (9) for inclusion in the bowel diary. Finally, a patient consultation meeting and a consensus meeting will be held for the participants who completed the Delphi survey.
Assessment of content validity of the newly developed bowel diary in a post-Delphi patient focus group consisting of 8-12 participants | 12 months
  Content validation of the newly developed bowel diary will be tested during interview in the post-Delphi patient focus group. This focus group is recorded using an audio and video recording. This recording are transcribed verbatim by the researcher into a Word document. The transcription will be analyzed using NVIVO 9 software.
The usability of the newly developed e-diary, assessed with the System Usability Scale (SUS) in patients after rectal surgery for rectal cancer | 12 months
  The participants will be asked to use a newly developed electronic bowel diary for 7 consecutive days. This bowel diary will be available on the smartphone in the form of an application. After 7 days, the usability of this e-diary will be assessed with the System Usability Scale (SUS). The SUS is a questionnaire consisting of 10 items, utilizing a 5-point Likert scale to measure users' perceived satisfaction with the system. It includes two subscales focusing on usability and learnability. Scores on the SUS range from 0 to 100, with no direct correlation to percentiles (i.e., a score of 60 does not signify a usability level of 60%). Instead, a score of 70 points or higher is commonly employed as an initial threshold indicating acceptable usability. This benchmark is derived from the overall mean of more than 200 studies covering various systems and products.
The usability of the newly developed e-diary will be evaluated through conversations with patients who have undergone rectal surgery for rectal cancer, after these patients have used the e-diary for seven consecutive days | 12 months
  Participants will be instructed to use a newly developed electronic bowel diary via a smartphone app for seven consecutive days. The research will then conduct conversations with the participants covering aspects such as complexity, the need for additional support, application coherence, user-friendliness, pre-existing knowledge requirements, and suggestions for improvement. Audio and video recordings of these conversations will be transferred to the researcher's computer and subsequently transcribed into a Word document. The transcriptions will be analyzed using NVIVO 9 software.
Construct validity of the newly developed bowel e-diary: Known groups method | 12 months
  Patients will be divided into two groups based on their LARS score: no/minor LARS and major LARS. Over a 7-day period, patients will be asked to complete the bowel diary, which will then be examined to determine if there is a meaningful difference between the two groups. The Mann-Whitney U-test will be used to assess whether the difference is significant, and the C-index will be calculated to evaluate how well the test distinguishes between the groups. A C-index of 0.65 or higher would indicate that the test is effective at differentiating between the groups.
Construct validity of the newly developed bowel e-diary: Convergent and divergent validity | 12 months
  The bowel diary will be completed by patients over a 7-day period, while the questionnaires (such as LARS, MSKCC-BFI, COREFO, PAC-SYM, QLQ-C30) will be filled out on day 7.
  The correlation between the bowel diary and the questionnaires (such as LARS, MSKCC-BFI, COREFO, PAC-SYM, QLQ-C30) will be calculated. The correlation will be performed across the entire set of questionnaires and bowel diary items, while pairwise correlations at the subscale level will analyze the relationship between related factors.
Test-retest reliability of the newly developed bowel e-diary | 12 months
  To investigate the test-retest reliability of the newly developed bowel e-diary, patients will have to fill out the bowel diary application twice, each time for a continuous period of 7 days, during a period when the disorder and treatment do not change (i.e., after the end of adjuvant treatment and/or after closure of an eventual temporary postoperative ileostomy).
Responsiveness of the newly developed bowel e-diary in patients after rectal surgery for rectal cancer. The newly validated e-diary is the primary outcome. | 12 months
  To evaluate the responsiveness of the new bowel diary, patients will complete the diary for 14 consecutive days. The first 7 days (day 1-7) will be compared with the following 7 days (day 7-14). Internal responsiveness will be calculated using the Standardized Response Mean (SRM) for the bowel diary. External responsiveness will be assessed by calculating the SRM for both the bowel diary and the LARS score and MSKCC-BFI questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Geraerts, PhD, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided